CLINICAL TRIAL: NCT02136303
Title: Regional Kale as Source of Lutein and Zeaxanthin to Improve Vision of Patients With Age-related Macular Degeneration - an Alternative to Supplements With Isolated Xanthophylls
Brief Title: Regional Kale as Source of Lutein and Zeaxanthin to Improve Vision of AMD-patients
Acronym: KALESIGHT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Volker Boehm, PD Dr. Volker Böhm, University of Jena
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BO 1511/8-1
Record Dates: First submitted 2014-05-06; First posted 2014-05-13 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Changes in Macular Pigment Optical Density

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (14):
- S1-Placebo (Placebo Comparator): placebo capsule with all ingredients, but without active compound, intervention for 4 weeks, S1: Dosage-dependency
  Interventions: Dietary Supplement: S1: Dosage-dependency
- S1-1L (Experimental): capsule containing 1 mg lutein out of kale, intervention for 4 weeks, S1: Dosage-dependency
  Interventions: Dietary Supplement: S1: Dosage-dependency
- S1-2L (Experimental): capsule containing 2 mg lutein out of kale, intervention for 4 weeks, S1: Dosage-dependency
  Interventions: Dietary Supplement: S1: Dosage-dependency
- S1-5L (Experimental): capsule containing 5 mg lutein out of kale, intervention for 4 weeks, S1: Dosage-dependency
  Interventions: Dietary Supplement: S1: Dosage-dependency
- S2-Kale_extract (Experimental)
  Interventions: Other: S2: Kale extract versus kale purée
- S2-Kale_purée (Experimental)
  Interventions: Other: S2: Kale extract versus kale purée
- S3-Placebo (Placebo Comparator)
  Interventions: Other: S3: Kale extract: AMD-patients
- S3-AMD-Patients (Experimental)
  Interventions: Other: S3: Kale extract: AMD-patients
- S3-non-AMD (Experimental)
  Interventions: Other: S3: Kale extract: AMD-patients
- S1-Placebo-Tagetes (Placebo Comparator): capsule containing all ingredients, but without active compound, intervention for 4 weeks, S1: Dosage-dependency
  Interventions: Dietary Supplement: S1: Dosage-dependency
- S1-1L-Tagetes (Experimental): capsule containing 1 mg lutein out of tagetes, intervention for 4 weeks, S1: Dosage-dependency
  Interventions: Dietary Supplement: S1: Dosage-dependency
- S1-2L-Tagetes (Experimental): capsule containing 2 mg lutein out of tagetes, intervention for 4 weeks, S1: Dosage-dependency
  Interventions: Dietary Supplement: S1: Dosage-dependency
- S1-5L-Tagetes (Experimental): capsule containing 5 mg lutein out of tagetes, intervention for 4 weeks, S1: Dosage-dependency
  Interventions: Dietary Supplement: S1: Dosage-dependency
- S1-10L-Tagetes (Experimental): capsule containing 10 mg lutein out of tagetes, intervention for 4 weeks, S1: Dosage-dependency
  Interventions: Dietary Supplement: S1: Dosage-dependency

INTERVENTIONS:
Dietary Supplement: S1: Dosage-dependency — kale extract: placebo, 1 mg lutein, 2 mg lutein, 5 mg lutein tagetes extract: placebo, 1 mg lutein, 2 mg lutein, 5 mg lutein, 10 mg lutein
  Arms: S1-10L-Tagetes; S1-1L; S1-1L-Tagetes; S1-2L; S1-2L-Tagetes; S1-5L; S1-5L-Tagetes; S1-Placebo; S1-Placebo-Tagetes
Other: S2: Kale extract versus kale purée
  Arms: S2-Kale_extract; S2-Kale_purée
Other: S3: Kale extract: AMD-patients
  Arms: S3-AMD-Patients; S3-Placebo; S3-non-AMD

SUMMARY:
The age-related macular degeneration (AMD) is an age-dependent, multi-factorial disease. In Western industrial countries, it is the main cause of visual impairments. In Germany, approximately 4.5 million people suffer from AMD. Genetic as well as nutritional aspects are mainly important in AMD development. Until now, AMD-patients are advised to use supplements based on the carotenoids lutein and zeaxanthin, comprised in high doses and in isolated form. Results showing the effects of food items (kale, spinach) rich in lutein on improvement of vision are scarce. And how much is needed within the diet? Within the planned project, human intervention studies will investigate whether an oil-based kale extract or fresh kale can be used to improve vision of AMD-patients and persons aged 50+ (without AMD). The first study will use volunteers without AMD (>18 y) to investigate if there is a dose-dependent effect of lutein and zeaxanthin (out of a kale extract) on macular pigment optical density (MPOD). This study will also compare the bioavailability of the carotenoids from the extract and from a supplement. A second study (also using volunteers without AMD, >18 y) will compare the bioavailability of lutein and zeaxanthin from the extract and from kale purée. The third study will investigate the effect of the oil-based kale extract on improvements of MPOD and vision of AMD-patients and of a control group (volunteers 50+ without AMD).

Usually, the intestinal absorption of lutein and zeaxanthin is determined by analyzing changes in concentrations in blood plasma. A fast, non-invasive sampling will be evaluated to check the efficacy of an increased uptake of lutein. Thus, the project will test the usability of buccal mucosa cells to detect metabolic changes after an uptake of carotenoids. Besides, the determination of carotenoid contents in skin will be checked on its use as biomarker of carotenoids in plasma and macula.

Thus, the planned research project will evaluate two non-invasive markers of exposition on their usability as markers of absorption of lutein and zeaxanthin in blood and macula. In addition, the minimally needed dosage of lutein and zeaxanthin for AMD prevention will be determined to reduce the possible risk of currently recommended doses of these compounds. The project will also present alternatives (kale extract, kale purée) for AMD prevention and to improve vision to be used instead of currently used high-dose supplements.

ELIGIBILITY:
Inclusion Criteria:

* healthy, > 18 years, written consent

Exclusion Criteria:

* uptake of dietary supplements, glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
changes in macular pigment optical density MPOD [ODU: optical density units] | baseline and after 4/8 weeks, baseline and after 6/12/18/24 weeks
  Changes from baseline to various time points for different parameters of MPOD will be measured: changes in mean MPOD [ODU], changes in max. MPOD [ODU], changes in volume of MPOD [ODU x (degree)2], changes in area of MPOD [degree2]

CONTACTS AND LOCATIONS:
Locations (1):
- University Eye Hospital, Friedrich Schiller University Jena, Jena, Germany

REFERENCES:
- [Result] Arnold C, Winter L, Frohlich K, Jentsch S, Dawczynski J, Jahreis G, Bohm V. Macular xanthophylls and omega-3 long-chain polyunsaturated fatty acids in age-related macular degeneration: a randomized trial. JAMA Ophthalmol. 2013 May;131(5):564-72. doi: 10.1001/jamaophthalmol.2013.2851. PMID 23519529
- [Result] Arnold C, Jentsch S, Dawczynski J, Bohm V. Age-related macular degeneration: Effects of a short-term intervention with an oleaginous kale extract--a pilot study. Nutrition. 2013 Nov-Dec;29(11-12):1412-7. doi: 10.1016/j.nut.2013.05.012. PMID 24103519